CLINICAL TRIAL: NCT05649124
Title: The Effect of Acupressure on Perineal Pain Level in Primiparous Women With Episiotomy: A Randomized Controlled Study
Brief Title: Nonpharmacological Method for Relief of Episiotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, sena dilek, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: sdilek2
Record Dates: First submitted 2022-11-24; First posted 2022-12-13 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Pain
Keywords: Episiotomy, acupressure, pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Experimental): * Participants in this group will be interviewed at postpartum 3rd and 5th hours. The application will be explained and a voluntary consent form will be signed.
  * Participant Information Form will be filled in by the researcher by face-to-face interview.
  * The VAS and McGill Pain Questionnaire, which will be applied to evaluate perineal pain at the 3rd and 5th hours of the postpartum period, will be filled in by the participant.
  * In a total application where SP6, ST36 and LI4 points will be applied for 2 minutes, the total time will be 12 minutes.
  * After the application, the VAS and McGill Pain Questionnaire Evaluating Perineal Pain will be filled in by the participant.
  * The participant will be informed that the study has been completed.
  Interventions: Behavioral: Acupressure group
- Control group (No Intervention): * Participants in this group will be interviewed at postpartum 3rd and 5th hours. The application will be explained and a voluntary consent form will be signed.
  * Participant Information Form will be filled in by the researcher by face-to-face interview.
  * 3. VAS (Visual analog scale) and McGill Pain Questionnaire for Evaluating Perineal Pain will be required at 5th and 5th hours.
  * No application will be made other than routine applications.

INTERVENTIONS:
Behavioral: Acupressure group — A suitable environment will be prepared for mothers in terms of warmth and light, where privacy can be protected. The application points will be determined with the acu-point device by choosing the most comfortable position of the mother, leaving the application points open. The most preferred points LI4, SP6 and ST36 were selected among the points that were reported to be effective in relieving luterus pain by scanning the literature on the points to be compressed. Acupressure will be applied to the points (bidirectional, right and left) for 2 minutes, for a total of 8 minutes. Light pressure will be applied with the thumb of the practitioner's hand. Immediately after applying pressure for 2 minutes for each point, it is passed to the other point in the symmetrical region and the application is made without interruption. While practicing, the researcher will check the time using a digital wristwatch with a stopwatch.
  Arms: Acupressure group

SUMMARY:
The study is a randomized controlled study to evaluate the effectiveness of acupressure applied to primiparous pregnant women who underwent episiotomy in the early postpartum period.

The research was carried out between August 2022 and November 2022 at Düzce University Health Practice and Research Center with mothers who gave vaginal birth. The research was carried out with two groups as acupressure and control groups. The sample number was calculated using the G*Power 3.1.9.2 program and the acupressure group: 30 and the control group: 30. It was collected the research data with the Introductory Information Form and Visual Analog Scale. The participants in the acupressure group were interviewed at the 3rd and 5th hours after birth. The application announcement was made and they were allowed to sign the voluntary consent form. The VAS was filled by the participant before the application. Acupressure was applied to SP6, ST36 and LI4 points for a total of 12 minutes. After the application, the VAS was filled again by the participant.

No application was made to the control group. The data of the research was evaluated using the Statistical Package 22.0 program for Social Sciences. In the evaluation of the data; descriptive statistics was given as percentage, arithmetic mean±standard deviation, median and minimum-maximum values. Independent two-sample t-test was used for normally distributed variables and Mann-Whitney U test was used for non-normally distributed variables. Pearson Correlation test was applied to determine the relationship between the pain intensity of the acupressure group and the tests and to determine the relationship between the tests. Statistical significance level was accepted as p<0.05.

DETAILED DESCRIPTION:
Aim: This study was planned to examine the effect of acupuncture on perineal pain after episiotomy in the early postpartum period.

Research hypothesis:

H0: Acupressure application applied to pregnant women who underwent episiotomy in the postpartum period has no effect on reducing the level of perineal pain.

H1: Acupressure application applied to pregnant women who underwent episiotomy in the postpartum period reduces the level of perineal pain.

Type of Study: This study was designed as a randomized controlled experimental study.

Research Universe The population of the study consisted of participants who had vaginal birth, had episiotomy, and were primiparous , postpartum between the 3rd and 5th hours of the early postpartum period in Düzce University Health Practice and Research Center. The G- Power program was used to determine the sample of the study and it was planned to recruit a total of 60 participants ( 30 participants in the Acupressure group and 30 participants in the control group).

Random number generation program " Research " It will be determined from Randomizer's website and divided into two groups. Thus, the number of each mother and the group number were determined and recorded.

Research data "Participant Information Form, VAS (Visual Analog Scale ) for Evaluating perineal Pain )".

Exhibitor Information Form It was prepared by the researcher within the framework of the literature. The form consists of a total of 31 questions questioning women's socio -demographic, obstetric and perineal pain information. It is applied to postpartum women on the 1st day after delivery.

VAS (Visual analog scale) Evaluation of Perineal Pain The patient marks his or her pain on a 10 cm ruler with "no pain" at one end and the most severe pain at the other. The patient is told that there are two endpoints and to mark any place between these points appropriate to the severity of the pain. The distance between the onset of painlessness and this point marked by the patient is measured in centimeters and recorded. It is stated that VAS is more sensitive and reliable than other unidimensional scales in pain severity measurement . The VAS is more sensitive than the simple descriptive scale.

Application Procedure of the Study After obtaining the necessary permissions from the ethics committee and the institution for the implementation of the study, participants who had a vaginal delivery and met the inclusion criteria of the study were interviewed by the institution. Participants were informed that they could participate in the study without affecting the care received at the hospital and that they could leave the study at any time, and their voluntary consent was obtained. After the participants were included in the study, they were assigned to the study groups according to the electronic randomization table. The data were collected by face-to-face interviews by the researcher working in the delivery room of the hospital. VAS (Visual Analog Scale ) was filled in by the participants to evaluate postpartum perineal pain . The VAS (Visual analog scale), in which perineal pain was evaluated, was filled in by the participants in the postpartum acupressure group at the 3rd and 5th hours before and after the application. No application was made to the control group other than routine applications.

Acupressure Application Technique An environment where privacy can be protected and there are no external stimuli was prepared for the participants. The application started by leaving the application points open and choosing the most comfortable position for the participants. For this study, 3 points (6 points in total on both sides from each point) were determined and these points are SP6, the 6th point of the spleen meridian, LI4, the 4th point of the large intestine meridian , and ST36, the 36th point of the stomach meridian. In addition, expert opinion was taken to determine the points. The practitioner will respectively apply circular motions to the points and then apply pressure within two minutes. Although there is a difference in the order of use of the determined acupuncture points, this study was performed symmetrically to the LI4, SP6 and ST36 points, respectively. The practitioner will have a stopwatch to control the time.

Large Intestine Meridian Point 4 (He Gu /LI4):

Position: It is the point where the cambered muscle group is located when the thumb and index finger are brought closer together. In other words, it corresponds to the midpoint of the metacarpal bone of the index finger.

Application Technique: Press the point with thumb/middle finger in a circular or up and down direction along the meridian line for 2 minutes. Work on 2 points on both hands separately or simultaneously. Signs of the Spot: Although this area is often used for face, headache and toothache , it is also a frequently preferred area to increase alertness and reduce fatigue.

Indications: Although this area is generally used for face, head and toothache, it is also a frequently preferred area to increase alertness and reduce fatigue.

Spleen Meridian 6th Point ( Sanyinjiao /SP6):

Location: It is located on the inside of the shinbone, four fingers above the ankle.

Application Technique: Press the point with thumb/middle finger in a circular or up and down direction along the meridian line for 2 minutes. Work on 2 points on both legs separately or simultaneously.

Symptoms of the Point: This point, which is generally used for urological and pelvic problems, menstrual pain and insomnia, is also preferred in various studies to reduce fatigue.

Stomach Meridian 36th Point (ST36):

Location: It is located in the anterior part of the tibia, four fingers below the patella .

Application Technique: Press the point with thumb/middle finger in a circular or up and down direction along the meridian line for 2 minutes. Work on 2 points on both legs separately or simultaneously.

Spot Symptoms: Provides good digestive power and is effective in relieving constipation, diarrhea and bloating. It is a vital energy point in the prevention of diabetes, which can be caused by increased heartburn.

* Application to Acupressure Group

  * The participants in this group were interviewed at the 3rd and 5th hours after birth. The application was announced and the voluntary consent form was signed.
  * Participant Information Form was filled by the researcher through face-to-face interview.
  * The VAS to be applied to evaluate perineal pain at the 3rd and 5th hours after delivery was filled out by the participant.
  * The total duration of the application, in which SP6, ST36 and LI4 scores were applied for 2 minutes, was 12 minutes .
  * After the application, the VAS Perineal Pain Evaluation form was filled by the participant.
  * The participant was informed that the study was completed.
* Application to the Control Group

  * The participants in this group were interviewed at the 3rd and 5th hours after birth. The application was announced and the voluntary consent form was signed.
  * Participant Information Form was filled by the researcher through face-to-face interview.
  * 3. VAS (Visual analog scale) Evaluation of Perineal Pain was requested at 5th and 5th hours.
  * No application other than routine applications.

Statistical and Analytical Methods:

Statistical analysis will be performed using the IBM SPSS Statistic 22.0 (IBM Corp. , Armonk , NY, USA) program. Descriptive statistical methods (number, percentage, mean, standard deviation) will be used in the evaluation of sociodemographic data. Parametric tests (chi-square, T test, etc.) and non-paramedic tests (Mann-Whitney U Test, Kruskal Wallis, etc.) will be used in the comparison of categorical variables when it is seen that the data are suitable for normal distribution) will be used when it is not suitable for a normal distribution. P significance level will be accepted as 0.05 .

ELIGIBILITY:
Inclusion Criteria:

* Elementary school or higher education
* 18 years and over,
* Primiparous,
* Episiotomy was applied,
* Having a normal delivery in the hospital where the study was conducted,
* Able to speak and understand Turkish,
* No medical treatment to affect the pain,
* Perineal pain score is above 4 according to VAS (Visual analog scale),
* Participants who voluntarily agree to participate in the study will be included in the study.

Exclusion Criteria:

* Does not have sufficient mental health to fill out the questionnaire,
* Experiencing postpartum complications (bleeding, infection, etc.),
* With impaired tissue integrity in the area to be applied,
* Having genital infection
* Heir in perineum,
* Taking painkillers in the last 6 hours,
* Smoking or using alcohol
* Pharmacological and non-pharmacological intervention to reduce postpartum perineal pain,
* Excluding episiotomy in a different region of the perineum, In addition, those who want to leave the research at any stage of the research will be excluded from the research.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
VAS (Visual analog scale) Evaluation of Perineal Pain | It was applied to evaluate perineal pain just before the application of acupressure at the 3rd hours postpartum.
  The patient marks his or her own pain on a 10 cm ruler, which says no pain on one end and the most severe pain on the other end. The patient is told that there are two endpoints and to mark anywhere between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in pain severity measurement. The VAS is more sensitive than the simple descriptive scale.
VAS (Visual analog scale) Evaluation of Perineal Pain | It was applied to evaluate perineal pain just before the application of acupressure at the 5th hours postpartum.
  The patient marks his or her own pain on a 10 cm ruler, which says no pain on one end and the most severe pain on the other end. The patient is told that there are two endpoints and to mark anywhere between these points that matches the severity of the pain. The distance between the onset of no pain and this point marked by the patient is measured and recorded in centimeters. It is stated that VAS is more sensitive and reliable than other unidimensional scales in pain severity measurement. The VAS is more sensitive than the simple descriptive scale.

SECONDARY OUTCOMES:
VAS (Visual analog scale) Evaluation of Perineal Pain | It was applied to evaluate perineal pain immediately after acupressure application at the postpartum 3rd hour.
  The patient marks his or her own pain on a 10 cm ruler, which says no pain on one end
VAS (Visual analog scale) Evaluation of Perineal Pain | It was applied to evaluate perineal pain immediately after acupressure application at the postpartum 5th hour.
  The patient marks his or her own pain on a 10 cm ruler, which says no pain on one end

CONTACTS AND LOCATIONS:
Overall Officials: Sena Dilek Aksoy, Ph.D., Principal Investigator — Kocaeli University; Burcu Ozturk, M.Sc., Study Chair — Duzce Ataturk State Hospital
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No